CLINICAL TRIAL: NCT00626301
Title: Simplifying Antiretroviral Treatment in Virally Suppressed Children by Switching From Double Boosted Protease Inhibitors to Lopinavir/Ritonavir Monotherapy
Brief Title: Lopinavir/Ritonavir Monotherapy in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Khon Kaen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 077; IRB# 241/50
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: efficacy; safety; pharmacokinetics; LPV/r monotherapy; Thai children; efficacy safety LPV/r monotherapy maintenance; treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Children who have completed HIV-NAT 017. Children treated with other double boosted PIs such as indinavir plus lopinavir/ ritonavir are also included.
  Interventions: Drug: LPV/r

INTERVENTIONS:
Drug: LPV/r — LPV/r 230/57.5 mg/m2 orally q12h or the adjusted dose based on therapeutic drug monitoring of LPV/r prior to enrollment as maintenance monotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy (clinical, immunological, virological outcome), pharmacokinetics and safety of lopinavir/ritonavir (LPV/r) monotherapy maintenance in Thai children after viral load suppression with double boosted protease inhibitors (PIs).

DETAILED DESCRIPTION:
The commonly used antiretroviral (ARV) regimen in the Thai National Access to Antiretroviral Program for People Living with HIV/AIDS is non-nucleoside reverse transcriptase (NNRTI) based HAART. However, one of the most challenging concerns of antiretroviral therapy is the emergence of drug resistance mutants which occurs in 30-40% of treated patients. Children failing nucleoside reverse transcriptase inhibitor (NRTI)/NNRTI regimens have limited options for second line therapy especially in a developing country such as Thailand.

At HIV-NAT, the Thai Red Cross AIDS Research Centre, we had a trial using standard doses of double boosted PIs, Lopinavir/ritonavir and Saquinavir, HIV-NAT 017, in 50 HIV infected children who failed the first line regimen. This ongoing trial showed the good efficacy of the double boosted PI in children, significant increasing of CD4 and decreasing of HIV-RNA in children who adhered to the treatment. However, a high number of pill counts for this regimen, 5-8 pills every 12 hours, life long can affect adherence and treatment outcome. In the HIV-NAT 017 study, a 48 week intent to treat analysis, 38% and 50% of children had total cholesterol ≥ 200 mg/dl and triglycerides ≥ 150 mg/dl after double boosted PI. Those lipid levels were significantly elevated when compared to baseline (p < 0.001). Double boosted PIs are also very costly. Studies in adults have shown that double boosted PIs had a disadvantage in lipid effect compared to a single PI-based regimen.

Lopinavir/ritonavir, the only PI co-formulated with ritonavir, is recommended as a first-line option for antiretroviral-naive patients initiating PI-based therapy and has shown a high potency, efficacy, and safety in HIV patients with high genetic barriers to resistance. LPV/r has also shown excellent efficacy in ARV-experienced children.

Mono boosted PI therapy trials in HIV adults, as the maintenance therapy after suppressed viral load, have been shown to be effective and safe. This strategy not only decreases the number of pills per dose but also saves for ARV cost and might improve the patient's adherence. As maintenance monotherapy after HIV-1 viral suppression, lopinavir/ritonavir has shown efficacy in adult trials with 80-90% virological suppression. A pilot study of a switch to lopinavir/ritonavir (LPV/r) monotherapy from nonnucleoside reverse transcriptase inhibitor-based therapy was reported with 92% of the participants on treatment at week 48 having HIV RNA < 75 copies/mL.

Therefore, in this trial, we aim to see the efficacy and safety of lopinavir/ritonavir maintenance monotherapy in Thai HIV infected children after virological suppression from previous double boosted PIs.

By simplifying maintenance antiretroviral treatment in children who are virally suppressed from previous double boosted PIs to lopinavir/ritonavir monotherapy, we hope to achieve the following:

1. A decrease in total cholesterol, LDL and triglycerides
2. An improvement in quality of life and in adherence to ARVs
3. No change in viral load

ELIGIBILITY:
Inclusion Criteria:

1. HIV infected children ages 2 to 18 years
2. Treated with double boosted PIs during the last three months
3. Two consecutive plasma HIV-RNA levels < 50 copies/ml at least 3 months apart
4. Willing to restart HAART with the same regimen as before enrollment, when indicated
5. Signed written informed consent

Exclusion Criteria:

1. Active AIDS-defining disease at screening
2. Pregnancy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy (clinical, immunological, virological outcome), pharmacokinetics and safety of LPV/r monotherapy maintenance in Thai children after viral load suppression with double boosted PIs | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Praphan Phanuphak, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre; Pope Kosalaraksa, MD, Principal Investigator — Department of Pediatrics, Khon Kaen University
Locations (3):
- Thailand (3):
  - Department of Pediatrics, Chulalongkorn University Hospital, Bangkok, Bangkok
  - HIV-NAT, Bangkok, Bangkok
  - Department of Pediatrics, Khon Kaen University, Khon Kaen, Changwat Khon Kaen

REFERENCES:
- [Result] Bunupuradah T, Panthong A, Kosalaraksa P, Wongsabut J, Puthanakit T, Lumbiganon P, Chuanjaroen T, Sopharak C, Udompanit T, Prasitsuebsai W, Pancharoen C, Ananworanich J; HIV-NAT 077 Study Team. Simplifying antiretroviral therapy to lopinavir/ritonavir monotherapy did not improve quality of life and therapy adherence in pretreated HIV-infected children. AIDS Res Hum Retroviruses. 2014 Mar;30(3):260-5. doi: 10.1089/AID.2013.0204. Epub 2013 Dec 21. PMID 24274723
- [Result] Kosalaraksa P, Ananworanich J, Puthanakit T, Pinyakorn S, Lumbiganon P, Chuanjaroen T, Chobkarjing U, Phanuphak P, Pancharoen C, Bunupuradah T; HIV-NAT 077 Study Team. Long-term lopinavir/ritonavir monotherapy in HIV-infected children. Pediatr Infect Dis J. 2013 Apr;32(4):350-3. doi: 10.1097/INF.0b013e31827b1bd3. PMID 23190774
- [Result] Bunupuradah T, Kosalaraksa P, Puthanakit T, Mengthaisong T, Wongsabut J, Lumbiganon P, Phanuphak P, Burger D, Pancharoen C, Ananworanich J; HIV-NAT 077 Study Team. Monoboosted lopinavir/ritonavir as simplified second-line maintenance therapy in virologically suppressed children. AIDS. 2011 Jan 28;25(3):315-23. doi: 10.1097/QAD.0b013e32834231f5. PMID 21157298
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org